CLINICAL TRIAL: NCT05223673
Title: A Randomised, Open-label, Multi-centre, Two-arm Phase 3 Study Comparing Futuximab/Modotuximab in Combination With Trifluridine/Tipiracil to Trifluridine/Tipiracil Single Agent With a Safety Lead-In Part in Participants With KRAS/NRAS and BRAF Wild Type Metastatic Colorectal Cancer Previously Treated With Standard Treatment and Anti-EGFR Therapy
Brief Title: Phase 3 Study of Futuximab/Modotuximab in Combination With Trifluridine/Tipiracil Versus Trifluridine/Tipiracil Single Agent in Participants With Previously Treated Metastatic Colorectal Cancer
Acronym: COLSTAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to discontinue the study during the Lead-In part and the Phase III part was not started due to strategic reasons.
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL3-95026-001; 2021-003151-41 (EudraCT Number)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Futuximab/modotuximab; Trifluridine/tipiracil; Phase III; Safety Lead-In part; S95026; Sym004; Adult; Metastatic; Colorectal; Colorectal Cancer; EGFR
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — futuximab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Futuximab/modotuximab combined with trifluridine/tipiracil (Safety Lead-In and Phase III parts) (Experimental)
  Interventions: Biological: Futuximab/modotuximab; Drug: Trifluridine/Tipiracil
- Trifluridine/tipiracil (Phase III part) (Active Comparator)
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Biological: Futuximab/modotuximab — Concentrate for solution for infusion, futuximab/modotuximab will be administered via IV route, once weekly of each cycle at 9 mg/kg/dose at Cycle 1 Day 1 and then at 6 mg/kg/dose. Each cycle is up to 28 days.
  Arms: Futuximab/modotuximab combined with trifluridine/tipiracil (Safety Lead-In and Phase III parts)
Drug: Trifluridine/Tipiracil — Film-coated tablets of trifluridine/tipiracil (35 mg/m²/dose) will be administered orally before futuximab/ modotuximab administration, twice a day (BID) within 1 hour after completion of morning and evening meals, 5 days on/2 days off, over 14 days, followed by a 14-day rest. This treatment cycle will be repeated every 28 days.
  Arms: Futuximab/modotuximab combined with trifluridine/tipiracil (Safety Lead-In and Phase III parts)
Drug: Trifluridine/Tipiracil — Film-coated tablets of trifluridine/tipiracil (35 mg/m²/dose) will be administered orally twice a day (BID) within 1 hour after completion of morning and evening meals, 5 days on/2 days off, over 14 days, followed by a 14-day rest. This treatment cycle will be repeated every 28 days.
  Arms: Trifluridine/tipiracil (Phase III part)

SUMMARY:
This is a randomized phase III study with a safety lead-in part in patients with KRAS/ NRAS and BRAF Wild Type metastatic colorectal cancer who have previously received treatment with oxaliplatin, irinotecan, fluoropyrimidines, anti-VEGF agents and anti-EGFR antibodies. The main objective of the safety lead-in part is to assess safety and tolerability of futuximab/modotuximab in combination with trifluridine/tipiracil. The primary objective of the phase III part is to compare Overall Survival of futuximab/modotuximab in combination with trifluridine/tipiracil vs trifluridine/tipiracil monotherapy in patients with tumours that are KRAS/NRAS and BRAF wild-type (WT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of metastatic colorectal cancer (mCRC), not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumour without RAS (KRAS and NRAS) and BRAF V600E mutations based on Circulating tumour DNA (ctDNA) screening blood test analysis
* Participants with measurable or non-measurable lesion
* Participants must have received at least 2 prior regimens of standard chemotherapy for mCRC and had demonstrated progressive disease or intolerance to their last regimen
* Participants should have received previous treatment with commercially available anti-EGFR mAbs for ≥ 4 months
* Estimated life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate haematological, renal and hepatic function

Exclusion Criteria:

* Pregnancy, possibility of becoming pregnant during the study, breastfeeding woman
* Patients currently receiving or having received anticancer therapies within 4 weeks prior to the inclusion visit (Safety Lead-in part) or randomization visit (Phase 3 part).
* Major surgery within 4 weeks prior to the inclusion visit (Safety Lead-in part) or randomization visit (Phase 3 part) or participants who have not recovered from side effects of the surgery
* Participants with serious/active/uncontrolled infection
* Known clinically significant cardiovascular disease or condition
* Significant gastrointestinal abnormality
* Skin rash of Grade > 1 from prior anti-EGFR at the time of inclusion (Safety Lead-in part) or randomization (Phase 3 part), or any other skin toxicity precluding participation in the study according to investigator's discretion.
* Treatment with systemic immunosuppressive therapy within 4 weeks prior to inclusion (Safety Lead-in part) or randomization (Phase 3 part)
* Prior radiotherapy if completed less than 4 weeks before the inclusion visit (Safety Lead-in part) or randomization visit (Phase 3 part)
* Patients with other malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Ciardiello, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (15):
- United States (2):
  - University of Michigan Oncology Clinic | Rogel Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
- Belgium (3):
  - UZA Edegem, Edegem
  - UZ Leuven Campus Gasthuisberg, Leuven
  - CHUUCL Namur site Godinne, Yvoir
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herning Regional Hospital (Regionhospitalet Godstrup), Herning
  - Odense Universitetshospital, Odense
- Finland (2):
  - Docrates cancer center, Helsinki
  - TAYS (Tampere University Hospital), Tampere
- Hungary (4):
  - Magyar Honvédség Egészségügyi Központ Onkológiai Osztály, Budapest
  - Debreceni Egyetem, Klinikai Központ Onkológiai Klinika, Debrecen
  - Bács-Kiskun Megyei Kórház a Szegedi Tudományegyetem Általános Orvostudomáyi Kar Oktatókórháza, Kecskemét
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ Onkoterápiás Klinika, Szeged
- National Cancer Center Hospital East, Chiba, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  sponsored by Servier with a first patient enrolled as of 1 January 2004 onwards for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Ciardiello F, Yoshino T, Modest DP, Martin Fernandez L, Roby L, Fougeray R, Lockhart BP, Tabernero J. 436TiP COLSTAR: Randomized, open-label, multicentre, phase III study comparing futuximab/modotuximab plus trifluridine/tipiracil to trifluridine/tipiracil in KRAS/NRAS and BRAF wild type (wt) metastatic colorectal cancer (mCRC) previously treated with both standard and anti-EGFR treatment. Ann Oncol. 2022 Sep;33(Supplement 7):S733-S73. doi: 10.1016/j.annonc.2022.07.574
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sponsor decided to discontinue the study during the Lead-In part and the Phase III (randomized) part was not started due to strategic reasons.
Groups:
- Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts): Futuximab/modotuximab: Concentrate for solution for infusion, futuximab/modotuximab was administered via IV route, once weekly of each cycle at 9 mg/kg/dose at Cycle 1 Day 1 and then at 6 mg/kg/dose. Each cycle is up to 28 days.
  Trifluridine/Tipiracil: Film-coated tablets of trifluridine/tipiracil (35 mg/m²/dose) was administered orally before futuximab/ modotuximab administration, twice a day (BID) within 1 hour after completion of morning and evening meals, 5 days on/2 days off, over 14 days, followed by a 14-day rest. This treatment cycle was repeated every 28 days.
Period: Overall Study
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Started | 7
Completed | 0 (Study was terminated prior to completion)
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — Study termination | 6

BASELINE CHARACTERISTICS:
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6
  Race: Asian | 1
Primary tumour site [Count of Participants; unit: Participants]
  Rectosigmoid segment | 2
  Rectum | 4
  Sigmoid colon | 1
Site of metastasis [Count of Participants; unit: Participants]
  Liver | 5
  Lung | 6
  Distant lymph node | 3
  Bone | 1
  Other | 2
Disease duration (years) [Mean (Standard Deviation); unit: years] | 4.062 (2.630)
Time from first metastasis diagnosis to inclusion (months) [Mean (Standard Deviation); unit: months] | 37.784 (22.556)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) (Safety Lead-In Part)
Description: DLTs observed during a 28-day period. A DLT is defined as the following: A clinically significant AE graded according to the NCI-CTCAE version 5.0, observed during the initial 28- day treatment period following the first IMP administration. Assessed as unrelated to underlying disease, disease progression, intercurrent illness, or concomitant medications. At least possibly related to the IMPs (futuximab/modotuximab or trifluridine/tipiracil or both) by the investigator and meeting criteria as outlined in the protocol.
Time Frame: End of cycle 1 (Each cycle is up to 28 days)
Measure: Number; unit: dose-limiting toxicities (DLTs)
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 7
dose-limiting toxicities (DLTs) | 0

2. Primary Outcome: Overall Survival (OS) (In Double Negative, KRAS/NRAS and BRAF Wild Type Patients) (Phase III Part)
Description: Time elapsed from date of randomization until the date of death from any cause
Time Frame: up to 4 years 9 months
Population: Sponsor decided to discontinue the study during the Lead-In part and the Phase III part was not started due to strategic reasons. Therefore, outcome measure data is not available
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (Safety Lead-In Part)
Description: Time elapsed from the first IMP intake to death
Time Frame: up to 24 months
Population: No analysis done for this outcome measure as data was not collected.
Groups:
- Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts): Futuximab/modotuximab: Concentrate for solution for infusion, futuximab/modotuximab was administered via IV route, once weekly of each cycle at 9 mg/kg/dose at Cycle 1 Day 1 and then at 6 mg/kg/dose. Each cycle is up to 28 days.
  Trifluridine/Tipiracil: Film-coated tablets of trifluridine/tipiracil (35 mg/m²/dose) was administered orally before futuximab/ modotuximab administration, twice a day (BID) within 1 hour after completion of morning and evening meals, 5 days on/2 days off, over 14 days, followed by a 14-day rest. This treatment cycle was repeated every 28 days.
  The study was terminated during the safety lead-in part, prior to the start of the randomized part.
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (In Triple Negative) (Phase III Part)
Description: Time elapsed from the date of randomization into the study to disease progression/death
Time Frame: up to 4 years 9 months
Population: as for outcome 2
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival (Phase III Part)
Description: Time elapsed from the date of randomization into the study to disease progression/death
Time Frame: up to 4 years 9 months
Population: as for outcome 2
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 0

6. Secondary Outcome: Adverse Events (Phase III Part)
Description: Incidence, severity, and relationship of treatment emergent adverse event and treatment emergent serious adverse event
Time Frame: Through study completion, up to 4 years 9 months
Population: as for outcome 2
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Any AEs reported from the date of the first administration of IMP to 30 days after the last date of IMP administration (approximately 2 months)
Arm/Group | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts)
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts) (N=7)
Vertigo (Ear and labyrinth disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Futuximab/Modotuximab Combined With Trifluridine/Tipiracil (Safety Lead-In and Phase III Parts) (N=7)
Eosinophilia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Neutrophilia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Device related thrombosis (General disorders) | 1
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT05223673/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT05223673/SAP_001.pdf